CLINICAL TRIAL: NCT04027361
Title: Driving Performance in Patients Aged 18 to 25 Years With Attention-Deficit/Hyperactivity Disorder (ADHD) After a Single-Dose of Amphetamine Extended-Release Tablets: A Pilot, Double-Blind, Placebo-Controlled Study
Brief Title: Amphetamine Extended Release Tablets and Driving Performance in Subjects With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRI108-ADD-600
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amphetamine ER Tablets, 20 mg (Active Comparator): Double-blind amphetamine extended-release tablets, 20 mg dose, single tablet, administered at baseline
  Interventions: Drug: Amphetamine Extended Release (ER) Tablet 20 mg
- Placebo (Placebo Comparator): Matching double-blind placebo tablets, 20 mg dose, single tablet, administered at baseline
  Interventions: Drug: Amphetamine Extended Release (ER) Tablet 20 mg

INTERVENTIONS:
Drug: Amphetamine Extended Release (ER) Tablet 20 mg — A single 20 mg dose of amphetamine ER Tablet, orally administered
  Other Names: Amphetamine extended-release oral tablet 20 mg

SUMMARY:
The purpose of this study is to assess the effect on driving performance of a single dose of amphetamine extended-release tablets (20 mg/tablet) compared with placebo at 45 minutes and 10 hours post-dose in young adults with ADHD.

DETAILED DESCRIPTION:
At a single US-based study site, a driving simulation will be used to assess the effect on driving performance for the co-primary endpoints, study subjects' driving performance at 45 minutes and 10 hours post-dose, compared with placebo. Eligible subjects will be prescreened for ADHD but otherwise healthy, aged 18-25 years.

Driving simulations that simulate common driving events to which the study subject must react. The reactions to each event will be assessed. Using a parallel-group design, subjects will be assessed while on study drug, and while on placebo.

Safety assessments will include spontaneously reported treatment-emergent adverse events and vital signs at 4 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 25 years, inclusive, at the time of screening who have a valid driver's license.
2. Normal visual acuity (either uncorrected or corrected with glasses, contact lenses or surgery) at Screening based upon clinical assessment of the Investigator
3. Diagnosed with ADHD using the Diagnostic and Statistical Manual of Mental Disorders Version 5 (DSM-5) criteria based on ADHD module from the Mini-International Neuropsychiatric Interview (M.I.N.I) version 7.0.2.
4. IQ within normal range based upon clinical assessment of the Investigator.
5. For female participants, presently using an acceptable method of contraception based upon clinical assessment of the Investigator.
6. Willing to abstain from using any forms of cannabinoids (THC, CBD, hemp oil, etc.) for 2 weeks prior to the Driving Simulation Visit (if applicable).
7. Be able to understand, read, write, and speak English fluently to complete the study related materials.
8. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. Current or lifetime history of bipolar disorder or any psychotic disorder.
2. Current active symptoms of major depression generalized anxiety disorder, obsessive-compulsive disorder, panic disorder, or post-traumatic stress disorder based upon clinical assessment of the Investigator.
3. Known history of chronic medical illnesses including known structural cardiac disorders, serious cardiac conditions, serious arrhythmias, cardiomyopathy, and known family history of sudden death.
4. History of uncontrolled hypertension or a resting systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg. Patients with well-controlled hypertension on a stable dose for at least 3 months of anti-hypertensives will be allowed to participate.
5. Have clinically significant findings in vital signs measurements at Screening including:

   * Systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg (average of triplicate measurements)
   * Heart rate >100 bpm (average of triplicate measurements)
6. Known history or presence of significant renal or hepatic disease.
7. Use of monoamine oxidase inhibitors (MAOI), e.g. selegiline, tranylcypromine, isocarboxazid, phenelzine, linezolid, methylene blue, within 14 days of the Driving Simulator Visit.
8. Use of ADHD medications including all stimulants (methylphenidate, amphetamine or derivatives of any of these products), within 48 hours of the Driving Simulator Visit.
9. Participation in a clinical study in which an investigational drug was administered within 30 days prior to Screening.
10. Known history of allergy/hypersensitivity to amphetamine or any of the components of the test products.
11. Known history of lack of clinical response to amphetamine based upon Investigator assessment
12. Any uncontrolled medical condition that, in the opinion of Medical Monitor or Sponsor, would preclude study participation.
13. History or presence of alcohol dependence or substance abuse disorder or within the last 6 months based upon clinical assessment of the Investigator.
14. Positive urine pregnancy test at Driving Simulator Visit
15. Positive breath alcohol test at Driving Simulator Visit.
16. Patient's inability or unwillingness to follow directions from the study research staff.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Composite Reaction Time Score | Measured at pre-dose, 45 minutes and 3 hours post-dose
  Measurement of reaction time across a series of driving simulations

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States